CLINICAL TRIAL: NCT02482337
Title: Prospective Evaluation of Per-Oral Endoscopic Myotomy (POEM) of the Lower Esophageal Sphincter for the Treatment of Esophageal Swallowing Disorders
Brief Title: Per-Oral Endoscopic Myotomy for Esophageal Swallowing Disorders
Acronym: POEM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated by the Principal Investigator's to redesign it using more efficient processes.
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 014-103
Record Dates: First submitted 2015-05-07; First posted 2015-06-26 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- POEM procedure (Experimental): Patients who underwent POEM
  Interventions: Procedure: POEM

INTERVENTIONS:
Procedure: POEM — POEM procedure in the OR

SUMMARY:
The purpose of this study is to show that the Per-Oral Endoscopic Myotomy (POEM) procedure is an effective treatment for people with achalasia.

DETAILED DESCRIPTION:
Currently the most commonly performed definitive treatment for symptomatic esophago-gastric junction outflow obstruction is a laparoscopic esophageal myotomy (LEM). In this procedure the outer longitudinal and inner circular muscle fibers of the distal esophagus and proximal stomach are divided, releasing the spasm and resulting in an open lumen. Although this procedure is effective in relieving troubles swallowing and in improving esophageal emptying, it is often accompanied by the development of GERD (as the muscle division results in incompetence of the antireflux barrier, the lower esophageal sphincter). For this reason a laparoscopic esophageal myotomy is most often accompanied by a fundoplication, in which part of the fundus of the stomach is folded around the distal esophagus and sutured in place, recreating a flap-valve mechanism. (It is best to perform this at the time of the laparoscopic myotomy as reoperation in that area is difficult). The fundoplication however may be imperfect, and may result in some degree of outflow obstruction itself or fail to control reflux. LEM results in 80% to 90% global patient satisfaction; but 10-20% continue to experience moderate dysphagia and 10-35% will have GERD by esophageal pH testing.

Others have evaluated the possibility of surgically dividing the muscle fibers from within the esophagus, using an endoscope rather than a laparoscope, in an animal model. The first human experience was reported in Japan using a per-oral endoscope to (a) incise the mucosa in the proximal esophagus as an entry point, (b) create a submucosal tunnel downwards, (c) perform an esophageal myotomy of the distal esophageal circular muscle, and (d) close the mucosal entry site with clips. The creation of the submucosal tunnel for some distance before the myotomy is a safety measure, so that should the mucosal closure fail, native tissues will appose and help seal any leak (rather like the Z-entry for a thoracentesis). Subsequent to this initial report, multiple single-arm studies have reported that the technique is safe and is associated with excellent medium-term relief of dysphagia..

In the POEM technique no fundoplication is performed. By the endoscopic creation of an esophageal submucosal tunnel the inner circular muscle layer could be easily visualized and in contrast to conventional laparoscopic esophageal myotomy, the authors described the division of only this inner circular esophageal muscle layer leaving the outer longitudinal muscle layer intact. The distal esophagus is exposed in LEM, hence disrupting the attachments to the diaphragm. These attachments contribute to the overall antireflux mechanism. It is hypothesized that by only dividing the inner circular muscle, and not disrupting the contribution of the outer longitudinal muscle or the diaphragmatic attachments to the antireflux mechanism, POEM may not have the same potential for reflux as a LEM. If this is the case then an antireflux procedure may not be needed after the POEM procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient with symptomatic achalasia or EGJ outflow obstruction with a motility study, esophagram, and EGD consistent with EGJ outflow obstruction.
* Medical indication for surgical myotomy.
* Ability to undergo general anesthesia
* Age > 18 yrs. of age and <85 yrs. of age with ability to give informed consent
* Candidate for laparoscopic esophageal myotomy.

Exclusion Criteria:

* Previous chest radiotherapy.
* Eosinophilic esophagitis
* Barrett's esophagus
* Stricture of esophagus
* Malignant or premalignant esophageal lesion
* Contraindications for EGD.
* Unable to provide informed consent.
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-06; Primary Completion 2024-10 (Actual); Study Completion 2024-10 (Actual)

PRIMARY OUTCOMES:
Improvement in swallowing | 6 months after surgery
  Outcome measure will be assessed by a questionnaire based on the patient's ability to swallow, by radiographic study, upper gastrointestinal endoscopy and ambulatory reflux testing.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Leeds, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Pescarus R, Shlomovitz E, Swanstrom LL. Per-oral endoscopic myotomy (POEM) for esophageal achalasia. Curr Gastroenterol Rep. 2014 Jan;16(1):369. doi: 10.1007/s11894-013-0369-6. PMID 24362953
- [Background] Pasricha PJ, Hawari R, Ahmed I, Chen J, Cotton PB, Hawes RH, Kalloo AN, Kantsevoy SV, Gostout CJ. Submucosal endoscopic esophageal myotomy: a novel experimental approach for the treatment of achalasia. Endoscopy. 2007 Sep;39(9):761-4. doi: 10.1055/s-2007-966764. PMID 17703382
- [Background] Inoue H, Minami H, Satodate H, Kudo S. First clinical experience of submucosal endoscopic esophageal myotomy for esophageal achalasia with no skin incision. Gastrointestinal Endoscopy 69(5): AB122, 2009.
- [Background] Luketich JD, Fernando HC, Christie NA, Buenaventura PO, Keenan RJ, Ikramuddin S, Schauer PR. Outcomes after minimally invasive esophagomyotomy. Ann Thorac Surg. 2001 Dec;72(6):1909-12; discussion 1912-3. doi: 10.1016/s0003-4975(01)03127-7. PMID 11789770